CLINICAL TRIAL: NCT02932631
Title: EFFECTS OF CONSTRAINT-INDUCED MOVEMENT THERAPY Versus CONVENTIONAL PHYSICAL THERAPY ON FUNCTIONAL RECOVERY AND QUALITY OF LIFE AFTER STROKE
Brief Title: Different Methods of Physical Therapy for Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Larissa Salgado de Oliveira Rocha, researcher, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41597715.9.0000.5174
Record Dates: First submitted 2016-09-06; First posted 2016-10-13 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2016-10

CONDITIONS: Joint Loose Bodies
Keywords: hemiparesis; STROKE; neural plasticity; PHYSICAL THERAPY
MeSH Terms: conditions — Joint Loose Bodies; Paresis; Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONVENTIONAL PHYSICAL THERAPY group (Active Comparator): physical exercises divided into three phases:
  1. stretching, strengthening and/or mobilization;
  2. functional training of the affected muscles;
  3. functional training of the paretic limb.
  Interventions: Other: THERAPY CONTROL AND MOVEMENT OF INDUCTION
- containment therapy induced (Experimental): healthy side is restricted with splinting and exercises in hemiparetic member: carry out functional tasks individually. Each task will be held for 5 minutes, totaling 60 minutes of service
  Interventions: Other: THERAPY CONTROL AND MOVEMENT OF INDUCTION

INTERVENTIONS:
Other: THERAPY CONTROL AND MOVEMENT OF INDUCTION — Volunteers conventional physiotherapy group will stretching, strengthening and / or mobilization and functional training of the affected muscles with 3 sets of 10 repetitions for 60 minutes.
  The restriction therapy group and induction motion the volunteers will wear a brace on the top healthy member to be restricted in each session during the exercises for this group for a period of 60 minutes, encouraging tasks involving activities of daily living and / or daily. In group practice mental, the volunteers listen to a CD that in the first two minutes, will promote progressive relaxation where imaginary in a calm and quiet place followed by 13 minutes of listening to the restriction therapy exercise protocol and motion induction. The association group practices and mental restriction therapy, volunteer listens to the CD for 15 minutes following the same procedures mentioned in group practice mental, followed by exercises functional activities for 45 minutes in the paretic limb.
  Other Names: PRACTICING MENTAL THERAPY; CONVENTIONAL PHYSICAL THERAPY

SUMMARY:
It is estimated that worldwide, about 15 million people are affected by vascular accident (CVA) per year, and in Brazil, the stroke is a major cause of death and disability, generating too much economic and social impact by generating motor sequelae , sensory and cognitive arising from blockage or rupture of blood vessels. Among the motor sequelae is the hemiparesis, which affects about 80% of cases with consequent impairment of the quality of life of individuals. However, physical therapy has shown to facilitate return of the function of these individuals, while minimizing the sensorimotor deficits for promoting neuronal plasticity through the motor relearning. Among the features of physical therapy are the conventional physical therapy techniques, Therapy and Restriction of Movement Induction (TRIM) and the Mental Practice. In view of this, the objective of the study is to compare the application of conventional physiotherapy protocols and TRIM and / or mental practice on the morphometric features, functionality and quality of life of post-stroke hemiparetic subjects in the chronic phase. 60 volunteers will be selected, of both sexes, aged between 45 and 80 years with a clinical diagnosis of stroke, with hemiparesis in the chronic phase were divided into four groups (N = 15): control group (CG), TRIM Group (GT), Mental Practice group (GPM) and group TRIM + Mental Practice (GTPM) to perform specific exercises for each group for three times a week, totaling 24 sessions. Volunteers will be evaluated in four times through the Fugl-Meyer Assessment scale (FMA) adapted and Motor Ability Test of the Upper Limb (THMMS) and to assess the Quality of Life will be used Quality Scale Specific Life Vascular Accident brainstem (EQVE-AVE) and oxidative stress analysis by collecting blood and electromyography for muscular activity. After the research data will be tabulated on an Excel spreadsheet to perform intergroup and intragroup comparisons between the four evaluation times, which will be used for data analysis the BioEstat® 5.2 program, the choice of tests for analysis dependent on the statistical distribution types found and the homogeneity of their variances.

DETAILED DESCRIPTION:
The sample is composed of 60 volunteers of both sexes, with a clinical diagnosis of stroke (CVA) with injury over six months time that characterizes the chronic stage of the disease and present hemiparesis in upper limb.

PROCEDURES AND DATA COLLECTION

The research will be divided into the following steps:

STAGE 1: The search will begin with an invitation to volunteers to participate in the study, through posters and verbal invitation. Then, a pre-selection candidates by applying MMSE will be performed, Jaeger card and Whisper test in order to evaluate the existence of cognitive impairment, visual and auditory respectively. If they can make up the sample, volunteers will be selected as meeting the inclusion and exclusion criteria, and researchers will deliver two-way the IC explaining how occur the research objectives of the Office and application of the Protocol and deliver two-way also statement of photographs and footage authorization for display permit photos and footage. It is noteworthy that both routes of the term and Declaration will be signed on every page by volunteers, which will be a copy of each document with the same.

Prior to the procedures and data collection, the researchers will be trained in the application of all instruments of evaluation and handling of resources to be used in the treatment of volunteers.

2nd STAGE: Volunteers will be evaluated through the scale application of FMA and THMMS in order to analyze the functionality and ability of MS and QOL will be assessed by EQVE-stroke as described in materials in this methodology.

The amplitude of the paretic upper limb movement will also be assessed by goniometry scapulohumeral humeral joint, shoulder, elbow, wrist, thumb interphalangeal and where use of a universal manual goniometer and another smaller toward the measuring fingers. The first measure goniometric be obtained after the patient's arrival in treatment- place in the pre-treatment. The following measures will be during treatment (12 ° session) and the immediate and late stages after the treatment. To perform such a procedure will be asked to volunteers who remain supine on a stretcher, followed by the sitting position in a chair, the latter should position the upper limb aligned to the trunk and forearm to be evaluated on a small table, a neutral pronation and supination with the elbow held in 90 ° of flexion.

3rd STAGE: Next muscle electromyographic activity will be measured by electromyography apparatus of Miotec ®.

Volunteers will conduct the test in a well-lit room with adequate ventilation and environment without noise, which will be placed in the sitting position with arm supported on fixed surface and so will surface electrodes connected on the paretic upper limb having as guidance for positioning electrodes muscular motor points previously located by an electrical stimulator and coupled with a conductive gel, so as to promote a more stable transitions and tendon insertions in order to quantitatively analyze the information sent nerve member.

The investigators will be asked to volunteer to perform three isometric contractions for four seconds each with two intervals between contractions two minutes, and asked each contraction the patient to reach its maximum strength. The muscles to be analyzed will be the flexors of fingers flexors wrist flexor ulnar elbow flexors, shoulder flexors and internal rotators of the shoulder, the answers will be measured and displayed on a computer screen that will be BIOPAC ® system.

4th STAGE: As for the functional range of the MS paretic will be measured by the functional reach test, adapted to the sitting position, in which the individual will be sitting without armrest in the chair for the upper limb, positioned laterally to the wall, with shoulder 15 cm away from this without touching it at any time, with feet parallel in a comfortable position, keeping the shoulder near the wall flexed to 90 °. A tape measure is fixed parallel to the floor, positioned at the height of the acromion. The volunteer will then be instructed to lean forward as much as possible; the displacement to be measured on the tape with three attempts functional range, then obtaining the average of the three.

5th STEP: Then, for the collection of handgrip strength in paretic MS will be used hydraulic dynamometer handgrip Jamar® where with volunteers in the sitting position in the bed, standing with the shoulder in neutral position, elbows and wrist in 90 ° neutral position, the therapist will support the dynamometer. Volunteers will be instructed to perform three handgrip maneuvers reaching maximum voluntary contraction with each hand, with one-minute interval between one operation and another. After the collection will be the simple arithmetic average entrees the three measures collected.

These procedures in the study will take place in four stages: before the start of treatment that correspond to the pre-treatment; after the 12th session that correspond to intermediate treatment; immediately after the 24th session, which will correspond to the immediate post-treatment; and the total intervention time equal to 24 sessions, which will be distributed in three weekly sessions held on alternate days (Monday, Wednesday and Friday). After evaluating the functionality evaluation of oxidative stress. Initially it will be collected blood with a sterile needle through the lancing on the medial side of the digital pulp of the fourth finger of the left hand, which will be pre-cleaned with 70% alcohol. The collection of blood drop will be made with a razor through five light taps of this blade with the drop microscopy. After this, at room temperature (23 ° C), the blade will be kept in place protected from contact with the blood of nine minutes for the realization of the collected blood clotting process. At the end of this period, the morphology of these clots is microscopically observed under a 40X magnification.

Morphological evaluation of oxidative stress in plasm blood be evaluated according to the test known as Optical Microscopy for cell analysis in vitro or HLB test, also known under the designation of Dry layer oxidative test, which will be referred to as microscopic morphology oxidative stress in plasm (EEW).

The EEW provides indirect information on to oxidative stress, among others, using the following grading system the percentage of the discontinuous area of clot present in microscope slide: grade I (normal oxidative stress rate, with total area of discontinuous extracellular matrix (ME) less than 10%), grade II (mild stress, with ME discontinuity area between 10 to 20%), grade III (moderate stress with ME discontinuity the area between 20 30%), grade IV (severe stress, with ME discontinuity area between 30 to 40%) and the grade V (very severe stress, with the ME discontinuity area above 40%).

The respective assigned qualitative graduation will be logged into a spreadsheet for further analysis statistics. As a measure of standardization, the observation of morphological patterns of different clots will be performed by one of the researchers associated with assessment by OxyScanner the so-called program developed and marketed by Aldea Global Soluciones® (SFA), which give a copy of the software.

This evaluation will be done in four stages, which will use throughout the process coats, disposable gloves and masks, and will be held by only one of the researchers, in order to avoid bias in the research.

ELIGIBILITY:
Inclusion Criteria:

* will be included in the study volunteers with stroke diagnosis for six months or more lesions.
* showing hemiparesis
* with at least 20 of passive extension handle and 10 for the fingers (TREVISAN; TRINTINAGLIA, 2010)
* who are aged between 45 and 80 years
* independent of race, color and cultural socioeconomic status, that are experiencing higher score to 24 points on the MMSE, which are not performing physical therapy at the time of the study and who agree and sign the consent form.

Exclusion Criteria:

* volunteers with a diagnosis of stroke at least six months
* stroke recurrence
* double hemiparesis
* hemiplegia, which present associated diseases
* uncontrolled hypertension according to the Brazilian Guidelines on Hypertension (systolic blood pressure (BP)> 90 and <140 diastolic pressure (DP )> 50 and <90) and heart rate (HR) 80-100 bpm
* respiratory rate (RR) from 18 to 20 rpm, with 36 temperature, diabetes, heart disease, apraxia, aphasia, that are experiencing pain and deformities upper limb, that are experiencing cognitive impairment, visual and hearing impairment, which will be assessed using the Mini Mental State Examination -MEEM tests (Appendix a) with scores below 24 points or taking into account score for illiterates, Jaeger Card (ANNEX B) and Test Whisper (ANNEX C) respectively
* who performs physical therapy at the time of the study, who do not agree and refuse to sign the Informed Consent

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
electromyography | pre-treatment and after 8 weeks
  For the evaluation of electrical muscle activity through electromyography through surface electrodes analyzed musculatures flexors and wrist extensors and elbow (median frequency, raw).
motor skills in the upper limbs | pre-treatment and after 8 weeks
  For evaluating the functionality of the Fugl-Meyer Assessment Scale was developed with the objective of evaluating six aspects of the patient, range of motion and pain, motor function, sensitivity, balance, coordination and speed. But the Motor Ability Test of the Upper Limb (THMMS) to measure quantitative and qualitative aspects of ADLs involving the upper limb in patients who have suffered strokes.Scales do not have measurement units only get a total points.
quality of life | pre-treatment and after 8 weeks
  Quality of Life Scale for Stroke (EQVE-AVE) which consists of 49 items, divided into 12 areas divided into energy, family role, language, mobility, humor, For the assessment of quality of life will be used Specific personality, self-care, social role, reasoning, upper limb function (MS), vision and work / productivity. Will be evaluated pre-treatment and after 24 sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Metodista de Piracicaba, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liepert J, Uhde I, Graf S, Leidner O, Weiller C. Motor cortex plasticity during forced-use therapy in stroke patients: a preliminary study. J Neurol. 2001 Apr;248(4):315-21. doi: 10.1007/s004150170207. PMID 11374097
- [Result] Jackson PL, Lafleur MF, Malouin F, Richards C, Doyon J. Potential role of mental practice using motor imagery in neurologic rehabilitation. Arch Phys Med Rehabil. 2001 Aug;82(8):1133-41. doi: 10.1053/apmr.2001.24286. PMID 11494195